CLINICAL TRIAL: NCT01127932
Title: Developing an Intervention to Address Suicide Risk During Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark A. Ilgen, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5R21DA026925-02 (NIH)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Suicide; Substance-Related Disorders
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Suicide; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT for suicide (Experimental)
  Interventions: Behavioral: CBT for suicide in Substance abuse
- Enhanced care control group (Active Comparator): This group is designed to be an active control which provides detailed information about substance use, suicide risk, and depression without providing any CBT or other specific therapy.
  Interventions: Behavioral: Psychoeducation for substance abuse

INTERVENTIONS:
Behavioral: Psychoeducation for substance abuse — This active control provides detailed information about substance use, suicide risk, and depression to those enrolled.
  Arms: Enhanced care control group
Behavioral: CBT for suicide in Substance abuse — The therapeutic intervention group is designed to provide beneficial coping strategies that are helpful in dealing with both substance use and suicidal thoughts.
  Arms: CBT for suicide

SUMMARY:
This is a 2-year study designed to: (1) adapt and refine an existing cognitive-behavioral treatment (CBT) intervention to decrease suicidal thoughts and behaviors for use in Substance Use Disorder (SUD) treatment settings, and (2) conduct a pilot randomized controlled trial with 50 patients in treatment for SUDs comparing the CBT intervention to an enhanced control condition. Through this pilot randomized controlled trial, the investigators hope to not only obtain information about the feasibility of implementing these procedures in residential SUD treatment, but to also determine whether this intervention decreases the level of suicidal ideation, suicide attempts, hopelessness, and frequency of substance use relative to the control condition.

DETAILED DESCRIPTION:
Existing research indicates that problematic alcohol and drug use are closely linked to both fatal and non-fatal suicide attempts. Given the strong association between substance use and suicide, an episode of substance use disorder (SUD) treatment provides a unique opportunity to decrease the likelihood of suicidal behaviors. However, there are no data on the effectiveness of specific interventions designed to decrease suicidal thoughts and behaviors during an episode of SUD treatment in individuals at high risk for suicide. Patients for this trial will be screened at the SUD treatment site for a combination of a past suicide attempt and current suicidal ideation and will be randomized to CBT or control conditions. All participants in the pilot randomized controlled trial will be assessed at baseline, at the end of treatment, and at a 3-month follow-up. From a public health perspective, SUD treatment programs contain large numbers of patients at high risk for future suicidal behaviors and therefore have the potential to play a central role in our nation's efforts to decrease suicide.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years of age
* Report a past lifetime suicide attempt
* Report current suicidal ideation
* Resided in treatment for less than 4 weeks
* In treatment for less than 6 months

Exclusion Criteria:

* Mental incompetence (e.g. unable to provide informed consent)
* Diagnosis of schizophrenia or currently psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Level of Suicidal Ideation | Six months

CONTACTS AND LOCATIONS:
Locations (1):
- Community Programs, INC., Waterford, Michigan, United States